CLINICAL TRIAL: NCT05852743
Title: Comparative Study Between Shear and Strain Elastography in Monitoring the Response to NAC in Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Silvia Gamal Rasmy, Resident doctor, Assiut University
Other Study IDs: SE and SWE in BC patients
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Monitoring the Response of Breast Cancer to Neoadjuvant Chemotherapy Using SE and SWE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: shear wave and strain elastography — shear wave elastography is a quantitative technique , while strain elastography is qualitative technique

SUMMARY:
The aim is to evaluate tumor stiffness changes through a comparative study between shear and strain elastography in monitoring the response of breast cancer to neoadjuvant chemotherapy

DETAILED DESCRIPTION:
Breast cancer (BC) is one of the most common malignant tumors in global population, with the highest morbidity and mortality rates among female.(1) Neoadjuvant chemotherapy (NAC) has become an important supplement of comprehensive and precise treatment of BC. Neoadjuvant chemotherapy (NAC) is increasingly used to induce tumor shrinkage, thereby allowing smaller surgical resection, eliminating clinically silent micro metastases, and providing prognostic information based on the extent of pathologic response(.2-4) Pathological complete response (pCR) is increasingly seen after neoadjuvant chemotherapy (NACT) for invasive breast cancer. Confident identification of pCR may lead to less radical breast surgery and to sentinel node biopsy rather than axillary clearance in women with pre-treatment positive nodes.(5)Response to NACT is routinely assessed using magnetic resonance imaging (MRI), greyscale ultrasound (US), and mammography.(6) In some studies, MRI has been shown to be superior to US.(7-8) however, MRI has the disadvantages of being time-consuming, expensive, requiring intravenous contrast agent . Ultrasonic elastography (UE) has been widely used to qualitatively and quantitatively evaluate differences in lesion stiffness or elasticity. Currently, the two most frequently used UE techniques for examination of breast diseases are strain elastography (SE) and shear-wave elastography (SWE). In practice, UE is a complementary technique for differentiating benign from malignant breast masses (9,10). Breast cancers with more aggressive pathological properties tend to have higher stiffness values .Strain elastography (SE) may be predictive of response in the early stage of treatment with high sensitivity (SEN) and specificity (SPE).(11,12) Pretreatment tumor stiffness measured by shear wave elastography (SWE) has a significant relationship with the subsequent reduction in tumor cellularity.(13) In case of NACT, early evaluation of relative changes in tumor stiffness could effectively predict the response and might indicate better therapeutic strategies.(14)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive ductal carcinoma .
2. Age equal or above 18

Exclusion Criteria:

1. Previous radiation therapy or chemotherapy
2. Mass not detected by US
3. Non Mass lesion by MRI
4. Ductal carcinoma in situ

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: a total of 65 female patient with biopsy confirmation of invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
comparative study between shear and strain elastography in monitoring the response of breast cancer to neoadjuvant chemotherapy | baseline
  evaluate tumor stiffness changes through a comparative study between shear and strain elastography in monitoring the response of breast cancer to neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Mohamed Refaat, Study Chair — Ass.Professor docotor ,diagnostic radiology department , in south egypt cancer institute; Shereen Ezzat Amin, Study Chair — lecturer doctor , diagnostic radiology department , in south egypt cancer institute; Eman Abo Elhamd, Study Chair — Professor doctor , diagnostic radiology department , assuit university